CLINICAL TRIAL: NCT02113878
Title: A Phase Ib Study of BKM120 With Weekly Cisplatin and Radiotherapy in High Risk Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Phase Ib Study of BKM120 With Cisplatin and XRT in High Risk Locally Advanced Squamous Cell Cancer of Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-008
Record Dates: First submitted 2014-04-01; First posted 2014-04-15 (Estimated); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Hypopharyngeal Cancer; Early Invasive Cervical Squamous Cell Carcinoma; Carcinoma of Larynx; Cancer of Nasopharynx
Keywords: Carcinoma, Squamous Cell of Head and Neck; Human Papillomavirus Positive Oropharyngeal Carcinoma; Hypopharyngeal Cancer; Early Invasive Cervical Squamous Cell Carcinoma; Carcinoma of Larynx; Cancer of Nasopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Neoplasms | interventions — NVP-BKM120; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Level 1 (Experimental): * 40 mg BKM120 will be administered orally daily for 45 days. Starting dose 40 mg.
  * Cisplatin: Starting Dose 30 mg/m2, given IV, weekly on days: (1, 8, 15, 22, 29, 36 and 43).
  * Radiotherapy: All participants will receive daily radiotherapy with intensity-modulated radiotherapy (IMRT) for 7 weeks.
  Interventions: Drug: BKM120; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy (IMRT)
- Dose Level 2 (Experimental): * 40 mg BKM120 will be administered orally daily for 45 days.
  * Cisplatin: Starting Dose 35 mg/m2, given IV, weekly on days: (1, 8, 15, 22, 29, 36 and 43).
  * Radiotherapy: All participants will receive daily radiotherapy with intensity-modulated radiotherapy (IMRT) for 7 weeks.
  Interventions: Drug: BKM120; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Drug: BKM120 — BKM120 is a potent and highly specific oral pan-class I PI3K inhibitor.
  Other Names: Buparlisib
Drug: Cisplatin — Cisplatin is a chemotherapy drug
  Other Names: Platinol-AQ; Platinol
Radiation: Intensity-modulated radiotherapy (IMRT) — IMRT is the medical use of ionizing radiation, generally as part of cancer treatment to control or kill malignant cells
  Other Names: IMRT

SUMMARY:
This research study is evaluating a drug called buparlisib (BKM120) as a possible treatment for locally advanced head and neck squamous cell cancer.

DETAILED DESCRIPTION:
* This phase Ib study is combining standard chemoradiotherapy with weekly cisplatin and BKM120 to assess tolerability of this combination in high risk patients with locally advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN). The investigators will also obtain preliminary information about the efficacy of this treatment.
* The participant will receive the study drug buparlisib once daily, by mouth, for 45 days. The participant will be given a study drug-dosing diary for each cycle. It will include special instructions for taking the study drug at home.
* The investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects, not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study before and how well they have tolerated their doses.
* All participants will receive weekly cisplatin injection. Cisplatin will be given intra-venously (IV) on days: (1, 8, 15, 22, 29, 36 and 43) at DFCI.
* All participants will receive daily radiotherapy with intensity-modulated radiotherapy (IMRT) for 7 weeks, delivered at DFCI. IMRT is a type of 3-dimensional radiation therapy that uses computer-generated images to show the size and shape of the tumor. Thin beams of radiation of different intensities are aimed at the tumor from many angles. This type of radiation therapy reduces the damage to healthy tissue near the tumor.
* The investigators would like to keep track of the participant's medical condition. Follow-up will continue every 4 to 12 weeks after the end of treatment for the first year and at the investigator's discretion thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Stage III/IV, locally advanced, biopsy proven squamous cell cancer of the head and neck that undergo chemoradiation as their primary treatment with curative intent.
* Oropharynx (HPV positive and HPV negative), hypopharynx, larynx primaries, nasopharynx as well as those with documented SCC of the cervical lymph nodes, with unknown primaries.
* >10 pack years of tobacco use
* Age ≥ 18 years
* ECOG performance status ≤ 2
* At least one site of measurable disease
* Adequate bone marrow function as shown by: ANC > 1.5 x 109/L, Platelets >100 x 109/L, Hb >9 g/dL
* Total calcium (corrected for serum albumin) within normal limits
* Magnesium ≥ the lower limit of normal
* Potassium within normal limits for the institution.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range
* Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
* Serum amylase ≤ ULN
* Serum lipase ≤ ULN
* Fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
* Signed informed consent
* INR ≤ 2

Exclusion Criteria:

* Distant metastatic disease
* Less than or equal to 10 pack years of tobacco history
* Received prior chemotherapy
* Received prior radiation to the head and neck or adjacent anatomical site
* Received prior treatment with a P13K inhibitor.
* Known hypersensitivity to BKM120 or to its excipients
* Acute or chronic liver, renal disease or pancreatitis
* Mood disorders ≥ CTCAE grade 3
* Diarrhea ≥ CTCAE grade 2
* Active cardiac disease
* History of cardiac dysfunction including any of the following:
* Patient has poorly
* Impairment of gastrointestinal (GI) function
* Currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug.
* Chronic treatment with steroids or another immunosuppressive agent.
* Herbal medications and certain fruits within 7 days prior to starting study drug.
* Currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Appendix B for a list of prohibited inhibitors and inducers of CYP3A (Please note that co-treatment with weak inhibitors of CYP3A is allowed).
* Undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control.
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Hanna, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share the IPD. Cumulative data will be published however.

REFERENCES:
- [Derived] Glorieux M, Dok R, Nuyts S. The influence of PI3K inhibition on the radiotherapy response of head and neck cancer cells. Sci Rep. 2020 Oct 1;10(1):16208. doi: 10.1038/s41598-020-73249-z. PMID 33004905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 29, 2014-December 5, 2017
Groups:
- Dose Level 1: * 40 mg BKM120 will be administered orally daily for 45 days. Starting dose 40 mg.
  * Cisplatin: Starting Dose 30 mg/m2, given IV, weekly on days: (1, 8, 15, 22, 29, 36 and 43).
  * Radiotherapy: All participants will receive daily radiotherapy with intensity-modulated radiotherapy (IMRT) for 7 weeks.
  BKM120: BKM120 is a potent and highly specific oral pan-class I PI3K inhibitor.
  Cisplatin: Cisplatin is a chemotherapy drug
  Intensity-modulated radiotherapy (IMRT): IMRT is the medical use of ionizing radiation, generally as part of cancer treatment to control or kill malignant cells
- Dose Level 2: * 40 mg BKM120 will be administered orally daily for 45 days.
  * Cisplatin: Starting Dose 35 mg/m2, given IV, weekly on days: (1, 8, 15, 22, 29, 36 and 43).
  * Radiotherapy: All participants will receive daily radiotherapy with intensity-modulated radiotherapy (IMRT) for 7 weeks.
  BKM120: BKM120 is a potent and highly specific oral pan-class I PI3K inhibitor.
  Cisplatin: Cisplatin is a chemotherapy drug
  Intensity-modulated radiotherapy (IMRT): IMRT is the medical use of ionizing radiation, generally as part of cancer treatment to control or kill malignant cells
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 17 | 6
Completed | 14 | 6
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — patient non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 17 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.1) | 57.2 (4.17) | 62.0 (7.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 14 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 15 | 6 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 6 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Stage [Count of Participants; unit: Participants] — Either of the following indicate Stage 3:
  * It is at least 4 cm across, and no cancer cells are present in nearby structures, lymph nodes or distant sites.
  * It is any size but has not grown into nearby structures or distant sites. Cancer cells are present in one same-side lymph node and is at most 3 cm across.
  Any of the following indicate Stage 4:
  * Grown into nearby structures
  * Grown into deeper tissue
  * Has spread to multiple lymph nodes
  * Has spread to one lymph node and is either at least 3cm on the same side or at least 6cm on the opposite side.
  Participants
    Clinical Cancer Stage 3 | 0 | 2 | 2
    Clinical Cancer Stage 4 | 17 | 4 | 21
Primary Disease Site [Count of Participants; unit: Participants]
  Hypopharynx | 1 | 0 | 1
  Oral Cavity | 4 | 2 | 6
  Oropharynx | 11 | 1 | 12
  Larynx | 0 | 3 | 3
  Oth | 1 | 0 | 1
Smoking History [Count of Participants; unit: Participants]
  Yes | 17 | 6 | 23
  No | 0 | 0 | 0
Number of Pack Years [Count of Participants; unit: Participants]
  Greater than 10 | 17 | 5 | 22
  Less than or equal to 10 | 0 | 1 | 1
Current Smoker [Count of Participants; unit: Participants]
  Yes | 2 | 3 | 5
  No | 15 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Cisplatin
Description: The trial uses 3+3 design to determine maximum tolerated dose (MTD).
Time Frame: While on treatment, up to 66 days
Population: *One additional patient enrolled in Dose Level 1 per physician discretion
Measure: Number; unit: mg/m2
Groups:
- Dose Level 1 and Dose Level 2: * 40 mg BKM120 will be administered orally daily for 45 days.
  * Cisplatin: Starting Dose 30 mg/m2 (Dose Level 1) or 35 mg/m2 (Dose Level 2), given IV, weekly on days: (1, 8, 15, 22, 29, 36 and 43).
  * Radiotherapy: All participants will receive daily radiotherapy with intensity-modulated radiotherapy (IMRT) for 7 weeks.
  BKM120: BKM120 is a potent and highly specific oral pan-class I PI3K inhibitor.
  Cisplatin: Cisplatin is a chemotherapy drug
  Intensity-modulated radiotherapy (IMRT): IMRT is the medical use of ionizing radiation, generally as part of cancer treatment to control or kill malignant cells
Arm/Group | Dose Level 1 and Dose Level 2
Number analyzed (Participants) | 23
mg/m2 | 30

2. Secondary Outcome: Best Overall Response
Description: The best overall response for each patient is given per Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1) criteria:
  Complete Response (CR) - Disappearance of all target and non-target lesions and lymph node short axis is <10 mm and no new lesions
  Partial Response (PR)
  * Disappearance of target lesions and >=1 persisting non-target lesion or tumor marker levels above normal limits and no new lesions or
  * >=30% decrease in sum of target lesion diameter and no new lesions
  Stable Disease (SD)
  - Less than 5 mm increase in target lesion diameter unless it results in a >=20% increase in diameter and >=1 persisting non-target lesion or tumor marker levels above normal limits and no new lesions
  Progressive Disease (PD)
  * >20% increase in target lesion diameter, must be an absolute increase of 5mm or
  * Substantial worsening in non-target lesion or
  * New lesion present
Time Frame: Measured at end of treatment, up to 66 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 17 | 6
Participants
  Complete Response | 6 | 2
  Partial Response | 6 | 2
  Stable Disease | 0 | 1
  Progressive Disease | 3 | 0

3. Secondary Outcome: Median Time to Progression
Description: The median amount of time from baseline to progression and/or death. Patients known to be alive at last contact are censored at last contact. All patients alive at 24 months from baseline are censored at 24 months.
Time Frame: Up to 24 months (Progression is defined using RECIST v1.0 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 17 | 6
months | 14.5 [13.3 to 22.8] | NA [NA to NA] — Only 1 event occurred and 5 patients were censored. Therefor a median time to progression was not reached

4. Secondary Outcome: 24 Month Overall Survival
Description: The probability of survival at 24 months using Kaplan-Meier estimates. Patients alive at 2 years are censored at 2 years.
Time Frame: Up to 24 months
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 17 | 6
probability of survival | 0.929 [0.591 to 0.99] | 0.240 [0.239 to 0.246]

5. Secondary Outcome: Median Anxiety Score Change
Description: The median change in score on the Generalized Anxiety Disorder - 7 (GAD-7) questionnaire from baseline to cycle 9.GAD-7 has 7 questions and each question has score from 0 to 3. Sum score of all questions will be used as the final score. The final score ranges from 0 to 21. Higher score represents worse anxiety.
Time Frame: From baseline to cycle 9, up to 66 days.
Measure: Median (Full Range); unit: points
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 17 | 6
points | -0.5 [-5 to 6] | 0 [-3 to 1]

6. Secondary Outcome: Median Depression Score Change
Description: The median change in score on the Patient Health Questionnaire - 9 (PHQ-8) from baseline to cycle 9. PHQ-9 has 9 questions and each question has score from 0 to 3. Sum score of all questions will be used as the final score. The final score ranges from 0 to 27. Higher score represents worse depression.
Time Frame: From baseline to cycle 9, up to 66 days.
Measure: Median (Full Range); unit: points
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 17 | 6
points | 1 [-4 to 9] | 0 [-8 to 0]

7. Secondary Outcome: P13K Status by Response
Description: Phosphoinositide 3-kinase (PI3K) biomarker status, either positive or negative, analyzed using established methods from tumor biopsies. P13K status is reported by response, either responder (CR or PR) or non-responder (SD or PR).
Time Frame: Biopsies drawn up to 10 days from registration. Response measured at from baseline to cycle 9, up to 66 days.
Population: Biomarker data was not collected for all patients. Data reported for all patients who were biopsied.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 15 | 4
Participants
  P13K Positive - Responder | 2 | 1
  P13K Positive - Non-Responder | 1 | 1
  P13K Negative - Responder | 9 | 1
  P13K Negative - Non-Responder | 3 | 1

8. Primary Outcome: Maximum Tolerated Dose of BKM120
Description: The trial uses 3+3 design to determine maximum tolerated dose (MTD).
Time Frame: While on treatment, up to 66 days
Population: *One additional patient enrolled in Dose Level 1 per physician discretion
Measure: Number; unit: mg
Groups:
- Dose Level 1 and Dose Level 2: 40 mg BKM120 will be administered orally daily for 45 days. Cisplatin: Starting Dose 30 mg/m2 (Dose Level 1) or 35 mg/m2 (Dose Level 2), given IV, weekly on days: (1, 8, 15, 22, 29, 36 and 43).
  Radiotherapy: All participants will receive daily radiotherapy with intensity-modulated radiotherapy (IMRT) for 7 weeks.
  BKM120: BKM120 is a potent and highly specific oral pan-class I PI3K inhibitor. Cisplatin: Cisplatin is a chemotherapy drug Intensity-modulated radiotherapy (IMRT): IMRT is the medical use of ionizing radiation, generally as part of cancer treatment to control or kill malignant cells
Arm/Group | Dose Level 1 and Dose Level 2
Number analyzed (Participants) | 23
mg | 40

ADVERSE EVENTS:
Time Frame: Measured while on-treatment. From baseline to cycle nine, up to 66 days.
Description: All adverse events data were included in the serious adverse event table as no identifier to indicate SAE/OAE in the dataset, cannot separate them retrospectively.
Arm/Group | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 1/17 | 1/6
Serious Adverse Events (participants affected / at risk) | 17/17 | 6/6
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=17) | Dose Level 2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 12 | 6
Anxiety (Psychiatric disorders) | 4 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 2
Blurred vision (Eye disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Cholesterol high (Investigations) | 3 | 0
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Depression (Psychiatric disorders) | 5 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 10 | 6
Device related infection (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 3
Dizziness (Nervous system disorders) | 3 | 1
Dry eye (Eye disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 9 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 11 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 10 | 0
Dysphasia (Nervous system disorders) | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 3 | 0
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 1
Edema trunk (General disorders) | 2 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 9 | 5
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 1
Hallucinations (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 0
Hearing impaired (Ear and labyrinth disorders) | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 5 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 5 | 4
Insomnia (Psychiatric disorders) | 4 | 2
Investigations - Other, specify (Investigations) | 2 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Lip infection (Infections and infestations) | 1 | 1
Lipase increased (Investigations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphedema (Vascular disorders) | 8 | 2
Memory impairment (Nervous system disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 15 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 12 | 5
Neck edema (General disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 5 | 4
Pain (General disorders) | 3 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 2
Paresthesia (Nervous system disorders) | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Platelet count decreased (Investigations) | 7 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pustular (Infections and infestations) | 2 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Serum amylase increased (Investigations) | 2 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 1
Skin infection (Infections and infestations) | 2 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 2
Tooth discoloration (Gastrointestinal disorders) | 2 | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Weight loss (Investigations) | 2 | 6
White blood cell decreased (Investigations) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT02113878/Prot_SAP_000.pdf